CLINICAL TRIAL: NCT00992160
Title: A 28-Day, Polysomnographic and Subjective Assessment of Vestipitant (15mg/Day) for the Treatment of Primary Insomnia in Adult Outpatients
Brief Title: Vestipitant 28-day Tolerance Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 111364
Record Dates: First submitted 2009-07-16; First posted 2009-10-09 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Sleep Disorders
Keywords: Polysomnography (PSG); Adults; Primary Insomnia
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Initiation and Maintenance Disorders | interventions — vestipitant

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Active (Experimental): Vestipitant 15mg once daily
  Interventions: Drug: GW597599
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GW597599 — GW597599 15mg tablet
  Arms: Active
Drug: Placebo — Placebo to match GW597599 15mg tablet
  Arms: Placebo

SUMMARY:
This study is a 28-day polysomnographic and subjective assessment of oral Vestipitant 15mg/day for treatment of Primary Insomnia in adults outpatients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female aged 18-64 years inclusively with Diagnosis of Primary Insomnia according to Diagnostic and Statistical Manual of Mental Disorders -Text Revision (DSM-IV-TR) criteria 307.42
* PSG variables collected during 2consecutive PSG screening nights falling as follows: TST between 240-420 mins inclusive (both nights) - LPS (Latency to Persistent Sleep): mean not less than 20mins, each night not less than 15 mins - WASO (Wake After Sleep Onset): mean not less than 60mins, each night not less than 45mins
* Women: non child bearing potential or if child bearing potential agree on Contraceptive Methods listed in Protocol

Exclusion Criteria:

* clinically significant Psychiatric and neurological disorders (sleep disorders other than Primary Insomnia, history of alcohol orother substance abuse or dependnce);
* nightshift or rotating shift-work;
* Lifestyle habits in agreement with Protocol requirement: caffeine - alcohol intake and smoke
* healthy according to GSK criteria - laboratory and ECG limits set in the Protocol

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 161 (Actual)
Dates: Start 2009-05; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Nocturnal polysomngraphy | 6 weeks after start of treatment

SECONDARY OUTCOMES:
Subjective sleep assessments as performed by Post-Sleep Questionnaires and subject -rated Insomnia Severity Index | 4 weeks after start of treatment
Motor and cognitive functioning assessed by neurological tests (Romberg and Hee-to-toe) and Cognitive tests (Digit Symbol Substitution test and verbal Learning Memory test) | 4 weeks after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (7):
- Germany (7):
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Schwerin, Mecklenburg-Vorpommern
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Magdeburg, Saxony-Anhalt
  - GSK Investigational Site, Berlin, State of Berlin

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 111364 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register